CLINICAL TRIAL: NCT05206149
Title: Stimulation Test With Intranasal Glucagon for Corticotroph, Somatotroph and Antidiuretic Axes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Ezio Ghigo, Full Professor, A.O.U. Città della Salute e della Scienza
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: GST-intranasale
Record Dates: First submitted 2021-12-01; First posted 2022-01-25 (Actual); Last update posted 2022-01-25 (Actual); Status verified 2022-01

CONDITIONS: Hypopituitarism
MeSH Terms: conditions — Hypopituitarism

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal Administration of Glucagon (Experimental): Intranasal administration of glucagon in healthy subjects
  Interventions: Drug: Intranasal glugagon
- Intranasal Administration of Placebo (Placebo Comparator): Intranasal administration of placebo (isotonic saline solution) in healthy subjects
  Interventions: Drug: Intranasal placebo

INTERVENTIONS:
Drug: Intranasal glugagon — Intranasal glucagon is administered at the dose of 3 mg. This corresponds to the administration of a single dose of Baqsimi®.
  Other Names: Baqsimi®
  Arms: Intranasal Administration of Glucagon
Drug: Intranasal placebo — Intranasal placebo (represented by isotonic saline solution) is administered.
  Arms: Intranasal Administration of Placebo

SUMMARY:
The diagnosis of secondary hypoadrenalism and GH deficiency (GHD) often requires the performance of a dynamic test. The glucagon stimulation test (GST) is one of the options for evaluating hypothalamic-pituitary function, representing a stimulus for both the corticotropic and somatotropic axis, substantially safe and easily available. The standard procedure involves the intramuscular injection of 1-1.5 mg of glucagon based on the patient's weight.

In addition to its antero-pituitary function, glucagon has also shown its ability to stimulate neurohypophyseal secretion. Using the copeptin dosage, it has been shown that after the administration of glucagon in healthy subjects there is a significant release of ADH. However, the available data are scarse and there is no standardized protocol for the use of the glucagon test in diabetes insipidus.

At the moment, GST is not the most frequently chosen diagnostic option. In fact, despite having the advantage of being able to investigate different areas of anterohypophyseal and probably posterohypophyseal function at the same time, the test has some disadvantages: the prolonged duration makes the procedure challenging, the intramuscular injection can be unwelcome, and many variables can come into play in the definition of a normal response (age, BMI, glycemic status).

The recent introduction of a single-dose nasal powder formulation (Baqsimi®) could overcome some of the limitations of classic GST and make the procedure less demanding.

To date, no assessments are yet available regarding a purely diagnostic role in the context of hypopituitarism of this new formulation.

Through the knowledge of the physiological response of the adrenocortical, somatotropic and ADH axis to the administration of intranasal glucagon in healthy subjects, it will be possible to evaluate its possible application in the diagnosis of GH deficiency, central adrenal insufficiency and possibly diabetes insipidus.

ELIGIBILITY:
Inclusion Criteria:

- Any adult healthy subject (age >= 18 years old) and not meeting the exclusion criteria listed below

Exclusion Criteria:

* BMI < 18.5 kg/m2 or > 25 kg/m2
* Any active pharmacological treatment
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Change in serum ACTH levels between baseline and 15 minutes after glucagon/placebo administration | From baseline (0 minutes) to 15 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum ACTH (ng/L) at baseline (0 minutes) and after 15 minutes from glucagon/placebo administration.
Change in serum ACTH levels between baseline and 30 minutes after glucagon/placebo administration | From baseline (0 minutes) to 30 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum ACTH (ng/L) at baseline (0 minutes) and after 30 minutes from glucagon/placebo administration.
Change in serum ACTH levels between baseline and 45 minutes after glucagon/placebo administration | From baseline (0 minutes) to 45 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum ACTH (ng/L) at baseline (0 minutes) and after 45 minutes from glucagon/placebo administration.
Change in serum ACTH levels between baseline and 60 minutes after glucagon/placebo administration | From baseline (0 minutes) to 60 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum ACTH (ng/L) at baseline (0 minutes) and after 60 minutes from glucagon/placebo administration.
Change in serum ACTH levels between baseline and 75 minutes after glucagon/placebo administration | From baseline (0 minutes) to 75 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum ACTH (ng/L) at baseline (0 minutes) and after 75 minutes from glucagon/placebo administration.
Change in serum ACTH levels between baseline and 90 minutes after glucagon/placebo administration | From baseline (0 minutes) to 90 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum ACTH (ng/L) at baseline (0 minutes) and after 90 minutes from glucagon/placebo administration.
Change in serum ACTH levels between baseline and 120 minutes after glucagon/placebo administration | From baseline (0 minutes) to 120 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum ACTH (ng/L) at baseline (0 minutes) and after 120 minutes from glucagon/placebo administration.
Change in serum ACTH levels between baseline and 150 minutes after glucagon/placebo administration | From baseline (0 minutes) to 150 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum ACTH (ng/L) at baseline (0 minutes) and after 150 minutes from glucagon/placebo administration.
Change in serum ACTH levels between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum ACTH (ng/L) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in serum cortisol levels between baseline and 15 minutes after glucagon/placebo administration | From baseline (0 minutes) to 15 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum cortisol (µg/L) at baseline (0 minutes) and after 15 minutes from glucagon/placebo administration.
Change in serum cortisol levels between baseline and 30 minutes after glucagon/placebo administration | From baseline (0 minutes) to 30 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum cortisol (µg/L) at baseline (0 minutes) and after 30 minutes from glucagon/placebo administration.
Change in serum cortisol levels between baseline and 45 minutes after glucagon/placebo administration | From baseline (0 minutes) to 45 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum cortisol (µg/L) at baseline (0 minutes) and after 45 minutes from glucagon/placebo administration.
Change in serum cortisol levels between baseline and 60 minutes after glucagon/placebo administration | From baseline (0 minutes) to 60 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum cortisol (µg/L) at baseline (0 minutes) and after 60 minutes from glucagon/placebo administration.
Change in serum cortisol levels between baseline and 75 minutes after glucagon/placebo administration | From baseline (0 minutes) to 75 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum cortisol (µg/L) at baseline (0 minutes) and after 75 minutes from glucagon/placebo administration.
Change in serum cortisol levels between baseline and 90 minutes after glucagon/placebo administration | From baseline (0 minutes) to 90 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum cortisol (µg/L) at baseline (0 minutes) and after 90 minutes from glucagon/placebo administration.
Change in serum cortisol levels between baseline and 120 minutes after glucagon/placebo administration | From baseline (0 minutes) to 120 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum cortisol (µg/L) at baseline (0 minutes) and after 120 minutes from glucagon/placebo administration.
Change in serum cortisol levels between baseline and 150 minutes after glucagon/placebo administration | From baseline (0 minutes) to 150 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum cortisol (µg/L) at baseline (0 minutes) and after 150 minutes from glucagon/placebo administration.
Change in serum cortisol levels between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response of the corticotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum cortisol (µg/L) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in serum GH levels between baseline and 15 minutes after glucagon/placebo administration | From baseline (0 minutes) to 15 minutes after glucagon/placebo administration
  The response of the somatotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum GH (µg/L) at baseline (0 minutes) and after 15 minutes from glucagon/placebo administration.
Change in serum GH levels between baseline and 30 minutes after glucagon/placebo administration | From baseline (0 minutes) to 30 minutes after glucagon/placebo administration
  The response of the somatotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum GH (µg/L) at baseline (0 minutes) and after 30 minutes from glucagon/placebo administration.
Change in serum GH levels between baseline and 45 minutes after glucagon/placebo administration | From baseline (0 minutes) to 45 minutes after glucagon/placebo administration
  The response of the somatotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum GH (µg/L) at baseline (0 minutes) and after 45 minutes from glucagon/placebo administration.
Change in serum GH levels between baseline and 60 minutes after glucagon/placebo administration | From baseline (0 minutes) to 60 minutes after glucagon/placebo administration
  The response of the somatotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum GH (µg/L) at baseline (0 minutes) and after 60 minutes from glucagon/placebo administration.
Change in serum GH levels between baseline and 75 minutes after glucagon/placebo administration | From baseline (0 minutes) to 75 minutes after glucagon/placebo administration
  The response of the somatotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum GH (µg/L) at baseline (0 minutes) and after 75 minutes from glucagon/placebo administration.
Change in serum GH levels between baseline and 90 minutes after glucagon/placebo administration | From baseline (0 minutes) to 90 minutes after glucagon/placebo administration
  The response of the somatotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum GH (µg/L) at baseline (0 minutes) and after 90 minutes from glucagon/placebo administration.
Change in serum GH levels between baseline and 120 minutes after glucagon/placebo administration | From baseline (0 minutes) to 120 minutes after glucagon/placebo administration
  The response of the somatotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum GH (µg/L) at baseline (0 minutes) and after 120 minutes from glucagon/placebo administration.
Change in serum GH levels between baseline and 150 minutes after glucagon/placebo administration | From baseline (0 minutes) to 150 minutes after glucagon/placebo administration
  The response of the somatotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum GH (µg/L) at baseline (0 minutes) and after 150 minutes from glucagon/placebo administration.
Change in serum GH levels between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response of the somatotroph axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring serum GH (µg/L) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in plasma copeptin levels between baseline and 15 minutes after glucagon/placebo administration | From baseline (0 minutes) to 15 minutes after glucagon/placebo administration
  The response of the antidiuretic axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 15 minutes from glucagon/placebo administration.
Change in plasma copeptin levels between baseline and 30 minutes after glucagon/placebo administration | From baseline (0 minutes) to 30 minutes after glucagon/placebo administration
  The response of the antidiuretic axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 30 minutes from glucagon/placebo administration.
Change in plasma copeptin levels between baseline and 45 minutes after glucagon/placebo administration | From baseline (0 minutes) to 45 minutes after glucagon/placebo administration
  The response of the antidiuretic axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 45 minutes from glucagon/placebo administration.
Change in plasma copeptin levels between baseline and 60 minutes after glucagon/placebo administration | From baseline (0 minutes) to 60 minutes after glucagon/placebo administration
  The response of the antidiuretic axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 60 minutes from glucagon/placebo administration.
Change in plasma copeptin levels between baseline and 75 minutes after glucagon/placebo administration | From baseline (0 minutes) to 75 minutes after glucagon/placebo administration
  The response of the antidiuretic axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 75 minutes from glucagon/placebo administration.
Change in plasma copeptin levels between baseline and 90 minutes after glucagon/placebo administration | From baseline (0 minutes) to 90 minutes after glucagon/placebo administration
  The response of the antidiuretic axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 90 minutes from glucagon/placebo administration.
Change in plasma copeptin levels between baseline and 120 minutes after glucagon/placebo administration | From baseline (0 minutes) to 120 minutes after glucagon/placebo administration
  The response of the antidiuretic axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 120 minutes from glucagon/placebo administration.
Change in plasma copeptin levels between baseline and 150 minutes after glucagon/placebo administration | From baseline (0 minutes) to 150 minutes after glucagon/placebo administration
  The response of the antidiuretic axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 150 minutes from glucagon/placebo administration.
Change in plasma copeptin levels between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response of the antidiuretic axis to the administration of intranasal glucagon, compared to placebo, was evaluated by measuring plasma copeptin (pmol/L) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.

SECONDARY OUTCOMES:
Change in serum sodium levels between baseline and 15 minutes after glucagon/placebo administration | From baseline (0 minutes) to 15 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 15 minutes from glucagon/placebo administration.
Change in serum sodium levels between baseline and 30 minutes after glucagon/placebo administration | From baseline (0 minutes) to 30 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 30 minutes from glucagon/placebo administration.
Change in serum sodium levels between baseline and 45 minutes after glucagon/placebo administration | From baseline (0 minutes) to 45 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 45 minutes from glucagon/placebo administration.
Change in serum sodium levels between baseline and 60 minutes after glucagon/placebo administration | From baseline (0 minutes) to 60 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 60 minutes from glucagon/placebo administration.
Change in serum sodium levels between baseline and 75 minutes after glucagon/placebo administration | From baseline (0 minutes) to 75 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 75 minutes from glucagon/placebo administration.
Change in serum sodium levels between baseline and 90 minutes after glucagon/placebo administration | From baseline (0 minutes) to 90 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 90 minutes from glucagon/placebo administration.
Change in serum sodium levels between baseline and 120 minutes after glucagon/placebo administration | From baseline (0 minutes) to 120 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 120 minutes from glucagon/placebo administration.
Change in serum sodium levels between baseline and 150 minutes after glucagon/placebo administration | From baseline (0 minutes) to 150 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 150 minutes from glucagon/placebo administration.
Change in serum sodium levels between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum sodium (mmol/L) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in serum potassium levels between baseline and 15 minutes after glucagon/placebo administration | From baseline (0 minutes) to 15 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum potassium (mmol/L) at baseline (0 minutes) and after 15 minutes from glucagon/placebo administration.
Change in serum potassium levels between baseline and 30 minutes after glucagon/placebo administration | From baseline (0 minutes) to 30 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum potassium (mmol/L) at baseline (0 minutes) and after 30 minutes from glucagon/placebo administration.
Change in serum potassium levels between baseline and 45 minutes after glucagon/placebo administration | From baseline (0 minutes) to 45 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum potassium (mmol/L) at baseline (0 minutes) and after 45 minutes from glucagon/placebo administration.
Change in serum potassium levels between baseline and 60 minutes after glucagon/placebo administration | From baseline (0 minutes) to 60 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum potassium (mmol/L) at baseline (0 minutes) and after 60 minutes from glucagon/placebo administration.
Change in serum potassium levels between baseline and 75 minutes after glucagon/placebo administration | From baseline (0 minutes) to 75 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum potassium (mmol/L) at baseline (0 minutes) and after 75 minutes from glucagon/placebo administration.
Change in serum potassium levels between baseline and 90 minutes after glucagon/placebo administration | From baseline (0 minutes) to 90 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum potassium (mmol/L) at baseline (0 minutes) and after 90 minutes from glucagon/placebo administration.
Change in serum potassium levels between baseline and 120 minutes after glucagon/placebo administration | From baseline (0 minutes) to 120 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum potassium (mmol/L) at baseline (0 minutes) and after 120 minutes from glucagon/placebo administration.
Change in serum potassium levels between baseline and 150 minutes after glucagon/placebo administration | From baseline (0 minutes) to 150 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum potassium (mmol/L) at baseline (0 minutes) and after 150 minutes from glucagon/placebo administration.
Change in serum potassium levels between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum potassium (mmol/L) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in plasma osmolality between baseline and 15 minutes after glucagon/placebo administration | From baseline (0 minutes) to 15 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma osmolality (mOsm/kg) at baseline (0 minutes) and after 15 minutes from glucagon/placebo administration.
Change in plasma osmolality between baseline and 30 minutes after glucagon/placebo administration | From baseline (0 minutes) to 30 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma osmolality (mOsm/kg) at baseline (0 minutes) and after 30 minutes from glucagon/placebo administration.
Change in plasma osmolality between baseline and 45 minutes after glucagon/placebo administration | From baseline (0 minutes) to 45 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma osmolality (mOsm/kg) at baseline (0 minutes) and after 45 minutes from glucagon/placebo administration.
Change in plasma osmolality between baseline and 60 minutes after glucagon/placebo administration | From baseline (0 minutes) to 60 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma osmolality (mOsm/kg) at baseline (0 minutes) and after 60 minutes from glucagon/placebo administration.
Change in plasma osmolality between baseline and 75 minutes after glucagon/placebo administration | From baseline (0 minutes) to 75 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma osmolality (mOsm/kg) at baseline (0 minutes) and after 75 minutes from glucagon/placebo administration.
Change in plasma osmolality between baseline and 90 minutes after glucagon/placebo administration | From baseline (0 minutes) to 90 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma osmolality (mOsm/kg) at baseline (0 minutes) and after 90 minutes from glucagon/placebo administration.
Change in plasma osmolality between baseline and 120 minutes after glucagon/placebo administration | From baseline (0 minutes) to 120 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma osmolality (mOsm/kg) at baseline (0 minutes) and after 120 minutes from glucagon/placebo administration.
Change in plasma osmolality between baseline and 150 minutes after glucagon/placebo administration | From baseline (0 minutes) to 150 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma osmolality (mOsm/kg) at baseline (0 minutes) and after 150 minutes from glucagon/placebo administration.
Change in plasma osmolality between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma osmolality (mOsm/kg) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in serum glucose levels between baseline and 15 minutes after glucagon/placebo administration | From baseline (0 minutes) to 15 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum glucose (mg/dl) at baseline (0 minutes) and after 15 minutes from glucagon/placebo administration.
Change in serum glucose levels between baseline and 30 minutes after glucagon/placebo administration | From baseline (0 minutes) to 30 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum glucose (mg/dl) at baseline (0 minutes) and after 30 minutes from glucagon/placebo administration.
Change in serum glucose levels between baseline and 45 minutes after glucagon/placebo administration | From baseline (0 minutes) to 45 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum glucose (mg/dl) at baseline (0 minutes) and after 45 minutes from glucagon/placebo administration.
Change in serum glucose levels between baseline and 60 minutes after glucagon/placebo administration | From baseline (0 minutes) to 60 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum glucose (mg/dl) at baseline (0 minutes) and after 60 minutes from glucagon/placebo administration.
Change in serum glucose levels between baseline and 75 minutes after glucagon/placebo administration | From baseline (0 minutes) to 75 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum glucose (mg/dl) at baseline (0 minutes) and after 75 minutes from glucagon/placebo administration.
Change in serum glucose levels between baseline and 90 minutes after glucagon/placebo administration | From baseline (0 minutes) to 90 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum glucose (mg/dl) at baseline (0 minutes) and after 90 minutes from glucagon/placebo administration.
Change in serum glucose levels between baseline and 120 minutes after glucagon/placebo administration | From baseline (0 minutes) to 120 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum glucose (mg/dl) at baseline (0 minutes) and after 120 minutes from glucagon/placebo administration.
Change in serum glucose levels between baseline and 150 minutes after glucagon/placebo administration | From baseline (0 minutes) to 150 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum glucose (mg/dl) at baseline (0 minutes) and after 150 minutes from glucagon/placebo administration.
Change in serum glucose levels between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring serum glucose (mg/dl) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in plasma insulin levels between baseline and 15 minutes after glucagon/placebo administration | From baseline (0 minutes) to 15 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma insulin (mU/L) at baseline (0 minutes) and after 15 minutes from glucagon/placebo administration.
Change in plasma insulin levels between baseline and 30 minutes after glucagon/placebo administration | From baseline (0 minutes) to 30 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma insulin (mU/L) at baseline (0 minutes) and after 30 minutes from glucagon/placebo administration.
Change in plasma insulin levels between baseline and 45 minutes after glucagon/placebo administration | From baseline (0 minutes) to 45 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma insulin (mU/L) at baseline (0 minutes) and after 45 minutes from glucagon/placebo administration.
Change in plasma insulin levels between baseline and 60 minutes after glucagon/placebo administration | From baseline (0 minutes) to 60 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma insulin (mU/L) at baseline (0 minutes) and after 60 minutes from glucagon/placebo administration.
Change in plasma insulin levels between baseline and 75 minutes after glucagon/placebo administration | From baseline (0 minutes) to 75 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma insulin (mU/L) at baseline (0 minutes) and after 75 minutes from glucagon/placebo administration.
Change in plasma insulin levels between baseline and 90 minutes after glucagon/placebo administration | From baseline (0 minutes) to 90 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma insulin (mU/L) at baseline (0 minutes) and after 90 minutes from glucagon/placebo administration.
Change in plasma insulin levels between baseline and 120 minutes after glucagon/placebo administration | From baseline (0 minutes) to 120 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma insulin (mU/L) at baseline (0 minutes) and after 120 minutes from glucagon/placebo administration.
Change in plasma insulin levels between baseline and 150 minutes after glucagon/placebo administration | From baseline (0 minutes) to 150 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma insulin (mU/L) at baseline (0 minutes) and after 150 minutes from glucagon/placebo administration.
Change in plasma insulin levels between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring plasma insulin (mU/L) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in urine sodium levels between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring urine sodium (mmol/L) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in urine potassium levels between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring urine potassium (mmol/L) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in urine creatinine levels between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring urine creatinine (mg/dl) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in urine osmolality between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of glycometabolic and hydro-electrolyte biochemical balance was evaluated by measuring urine osmolality (mOsm/kg) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in resistance at bioimpedance vector analysis between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of bioimpedance vector analysis (BIVA) was evaluated by measuring resistance (Ohm) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in reactance at bioimpedance vector analysis between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of bioimpedance vector analysis (BIVA) was evaluated by measuring reactance (Ohm) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.
Change in phase angle at bioimpedance vector analysis between baseline and 180 minutes after glucagon/placebo administration | From baseline (0 minutes) to 180 minutes after glucagon/placebo administration
  The response to the administration of intranasal glucagon, compared to placebo, in terms of bioimpedance vector analysis (BIVA) was evaluated by measuring phase angle (°) at baseline (0 minutes) and after 180 minutes from glucagon/placebo administration.

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Città della Salute e della Scienza, Turin, Piedmont, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boguszewski CL. Glucagon stimulation test: has its time come? Endocrine. 2017 Sep;57(3):361-363. doi: 10.1007/s12020-017-1356-8. Epub 2017 Jun 23. No abstract available. PMID 28646378
- [Background] Arvat E, Maccagno B, Ramunni J, Giordano R, Broglio F, Gianotti L, Maccario M, Camanni F, Ghigo E. Interaction between glucagon and hexarelin, a peptidyl GH secretagogue, on somatotroph and corticotroph secretion in humans. Eur J Endocrinol. 2000 Nov;143(5):601-6. doi: 10.1530/eje.0.1430601. PMID 11078983
- [Background] Berg C, Meinel T, Lahner H, Yuece A, Mann K, Petersenn S. Diagnostic utility of the glucagon stimulation test in comparison to the insulin tolerance test in patients following pituitary surgery. Eur J Endocrinol. 2010 Mar;162(3):477-82. doi: 10.1530/EJE-09-0824. Epub 2009 Dec 8. PMID 19996199
- [Background] Yuen KC, Biller BM, Katznelson L, Rhoads SA, Gurel MH, Chu O, Corazzini V, Spiller K, Gordon MB, Salvatori R, Cook DM. Clinical characteristics, timing of peak responses and safety aspects of two dosing regimens of the glucagon stimulation test in evaluating growth hormone and cortisol secretion in adults. Pituitary. 2013 Jun;16(2):220-30. doi: 10.1007/s11102-012-0407-7. PMID 22806554
- [Background] Giuffrida FM, Berger K, Monte L, Oliveira CH, Hoff AO, Maciel RM, Vieira JG. Relationship between GH response and glycemic fluctuations in the glucagon stimulation test. Growth Horm IGF Res. 2009 Feb;19(1):77-81. doi: 10.1016/j.ghir.2008.06.002. Epub 2008 Aug 3. PMID 18678516
- [Background] Dichtel LE, Yuen KC, Bredella MA, Gerweck AV, Russell BM, Riccio AD, Gurel MH, Sluss PM, Biller BM, Miller KK. Overweight/Obese adults with pituitary disorders require lower peak growth hormone cutoff values on glucagon stimulation testing to avoid overdiagnosis of growth hormone deficiency. J Clin Endocrinol Metab. 2014 Dec;99(12):4712-9. doi: 10.1210/jc.2014-2830. PMID 25210883
- [Background] Hamrahian AH, Yuen KC, Gordon MB, Pulaski-Liebert KJ, Bena J, Biller BM. Revised GH and cortisol cut-points for the glucagon stimulation test in the evaluation of GH and hypothalamic-pituitary-adrenal axes in adults: results from a prospective randomized multicenter study. Pituitary. 2016 Jun;19(3):332-41. doi: 10.1007/s11102-016-0712-7. PMID 26897383
- [Background] Lewandowski KC, Lewinski A, Skowronska-Jozwiak E, Stasiak M, Horzelski W, Brabant G. Copeptin under glucagon stimulation. Endocrine. 2016 May;52(2):344-51. doi: 10.1007/s12020-015-0783-7. Epub 2015 Nov 17. PMID 26578365
- [Background] Guzman CB, Dulude H, Piche C, Rufiange M, Sadoune AA, Rampakakis E, Carballo D, Triest M, Zhang MX, Zhang S, Tafreshi M, Sicard E. Effects of common cold and concomitant administration of nasal decongestant on the pharmacokinetics and pharmacodynamics of nasal glucagon in otherwise healthy participants: A randomized clinical trial. Diabetes Obes Metab. 2018 Mar;20(3):646-653. doi: 10.1111/dom.13134. Epub 2017 Nov 19. PMID 29053231
- [Background] Sherr JL, Ruedy KJ, Foster NC, Piche CA, Dulude H, Rickels MR, Tamborlane WV, Bethin KE, DiMeglio LA, Fox LA, Wadwa RP, Schatz DA, Nathan BM, Marcovina SM, Rampakakis E, Meng L, Beck RW; T1D Exchange Intranasal Glucagon Investigators. Glucagon Nasal Powder: A Promising Alternative to Intramuscular Glucagon in Youth With Type 1 Diabetes. Diabetes Care. 2016 Apr;39(4):555-62. doi: 10.2337/dc15-1606. Epub 2016 Feb 16. PMID 26884472